CLINICAL TRIAL: NCT00443365
Title: Should we Repair Ischemic Mitral Regurgitation?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Silesia (Other)
Collaborators: Ministry of Health, Poland (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6/252/35/3747
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2008-05

CONDITIONS: Coronary Disease; Mitral Valve Insufficiency
MeSH Terms: conditions — Coronary Disease; Mitral Valve Insufficiency | interventions — Mitral Valve Annuloplasty

ARMS (2):
- 1 (No Intervention): Coronary Artery Bypass Grafting with no Mitral Valve intervention
- 2 (Active Comparator): Coronary Artery Bypass Grafting + Mitral Annuloplasty
  Interventions: Procedure: Mitral valve repair

INTERVENTIONS:
Procedure: Mitral valve repair — mitral valve annuloplasty
  Arms: 2

SUMMARY:
The purpose of this study is to assess whether adding mitral valve repair to coronary artery bypass grafting improves outcome in patients with ischemic mitral regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Stable coronary artery disease
* Patient accepted for coronary artery bypass surgery
* Ischemic mitral regurgitation

Exclusion Criteria:

* Acute coronary syndrome within 30 days
* Organic valvular heart disease
* Need for other than CABG and mitral valve repair cardiac surgical procedure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: Marek A Deja, MD PhD, Principal Investigator — Medical University of Silesia
Locations (1):
- 2nd Dept of Cardiac Surgery, Medical University of Silesia, Katowice, Poland